## **Borderline Personality Disorder and Emotion Regulation**

Effects of emotion-focused vs. cognitive schema therapy interventions on emotion regulation deficits in borderline personality disorder - associations between clinical efficacy, brain network function and local glutamate/GABA metabolism

Ethiks approval 04.06.2018, last time edited

## **Assessments**

| | T0<br>Inclusion<br>Therapy beginning | T1<br>End of therapy | T3 follow-<br>up 1 | T4<br>follow-up 2 | |
|---|---|---|---|---|---|
| | Week 1* | Week 9** | 6 month after therapy | 1 year after<br>therapy | |
| | Diagnostic phase | Outcome (1) | Outcome (2) | Outcome (3) | |
| PF-TK (s) | Х | | Х | | |
| SEFP (c) | Х | Х | Х | Х | ,<br> |
| <u>PID-5</u> (s) | х | X | Х | Х | |
| BPDSI-IV (c) | х | X | X | Х | |
| <u>EHI</u> (s) | х | | | | - • Diagnostics |
| CTQ (s) | х | | | | • Inclusion/exclusion criteria |
| IDA-R | (X) | | | | |
| WAIS-IV | (X) | | | | |
| ERI (s) | Х | Х | Х | Х | Primary outcome |
| FSVV (s) | х | X | X | Х | |
| BSL-95 (s) | Х | Х | Х | Х | |
| IIP (s) | х | X | X | Х | Secondary outcome (BPD-specific) |
| SMI (s) | х | X | X | Х | (2) 2 Specime, |
| YSQ-S3r (s) | х | X | X | Х | |
| BDI II (s) | Х | Х | Х | Х | To control for occurence and change of |
| SCL-90-R (s) | х | X | X | Х | depressive and other psychiatric symptoms |
| | *questionnaire<br>survey in week 1 | **questionnaire<br>survey in week 9 | (c) clinician-administere<br>(s) self-rated<br>(x) if applicable | d | acpressive and other payamatre symptoms |
| DE.TV (c) | Patient Questionnaire | | | Reference: | |

| PF-TK (s) | Patient Questionnaire Day-Clinic Jena | |
|---|---|---|
| SEFP (c) | Levels of Personality Functioning Scale (LPFS) | Bender et al. (2011) |
| PID-5 (s) | Personality Inventory for DSM-5 (Criterion B) | Krueger (2012), Zimmermann et al. (2014) |
| BPDSI-IV (c) | Borderline Personality Disorder Severity Index – fourth version | Arntz et al. (2003), Kröger et al. (2013, 2016) |
| EHI | Edinburgh Handedness Inventory | Oldfield (1971) |
| CTQ (s) | Childhood Trauma Questionnaire | Bernstein et al. (2003); Klinitzke et al (2012) |
| IDA-R | structured guide for the integrated diagnosis of adult ADHD | Retz et al. (2012) |
| WAIS-IV | Wechsler Adult Intelligence Scale - fourth version | Wechsler (2008) |
| ERI (s) | Emotion Regulation Inventory | König et al. (2011) |
| FSVV (s) | Questionnaire concerning self-harming behavior (modified) | Reicherzer & Brandl (2011) |
| BSL-95 (s) | Borderline Symptom List (95 Items) | Bohus et al. (2001, 2007) |
| IIP-D (s) | Inventory of Interpersonal Problems | Horowitz et al. (1988, 2000) |
| SMI (s) | Schema Mode Inventory (118 item version) | Lobbestael et al (2010), Reiss et al. (2012), Young et al. (2007) |
| YSQ-s3r (s) | Young Schema Questionnaire (short version) | Kriston et al. (2013), Phillips et al. (2017), Young et al. (1994) |
| BDI-II (s) | Beck Depression Inventory-II | Beck et al. (1996), Hautzinger et al. (2006), Kühner et al. (2007) |
| SCL-90-R (s) | Symptom Checklist-90-Revised | Derogatis (1979), Franke (2002), Schauenbuerg & Strack (1999) |